CLINICAL TRIAL: NCT00523133
Title: Posttreatment Effects of Naltrexone
Brief Title: Research on Individualized Treatment for Alcoholism
Acronym: RITA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency); Brown University (Other); George Washington University (Other)
Organization: Indiana University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01AA012696-01A1 (NIH)
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2007-08-31 (Estimated); Status verified 2007-08

CONDITIONS: Alcohol Dependence
Keywords: alcoholism; naltrexone; motivational enhancement therapy
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: naltrexone — 50 mg naltrexone daily for 3 months
Drug: naltrexone — 50 mg of naltrexone daily for 6 months
Behavioral: Broad Spectrum Treatment — 8-14, one hour sessions over 6 months
Behavioral: Motivational Enhancement Treatment — 4, 20 minute sessions over 3 months

SUMMARY:
The purpose of this study was to compare the effects of two psychosocial treatments that differed in scope and intensity (Broad Spectrum Treatment and Motivational Enhancement Treatment) combined with 3 or 6 months of treatment with naltrexone on alcohol drinking behaviors in alcohol dependent patients.

ELIGIBILITY:
Inclusion Criteria:

* men and women between the ages of 21-65
* current DSM-IV diagnosis of alcohol dependence
* abstinent for a minimum of 3 and maximum of 21 days prior to treatment initiation
* able to participate in an 18-month outpatient study
* live within a one hour or less commute to Fairbanks
* fluent in English
* women of child-bearing potential must have a negative pregnancy test and use effective contraceptive methods.
* score as contemplators or greater on the Readiness For Change Scale

Exclusion Criteria:

* severe hepatic disease (gGGT, SGOT or other liver functions greater than 4 times normal)
* opiate use (for any reason) in the last 14 days or a history of opioid dependence in the past year
* pregnant or lactating females or those unwilling to use birth control
* inability, according to the opinion of the interviewer, to follow medication instructions and safety precautions
* comorbid substance dependence (but not abuse) diagnosis in the past 6 months, excluding nicotine or marijuana dependence
* concomitant use of medications intended to decrease drinking (e.g. disulfiram)
* meeting current DSM criteria for bipolar disorder, schizophrenia, bulimia/anorexia, dementia, major depression

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2000-09; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Percent Days Abstinent | 18 months

SECONDARY OUTCOMES:
Percent Heavy Drinking Days | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Dena Davidson, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- University Hospital, Psychiatry Outpatient Clinic, Indianapolis, Indiana, United States